CLINICAL TRIAL: NCT06848023
Title: Clinical Outcomes of Patients 60 Years of Age and Older: Reverse Total Shoulder Arthroplasty Versus Rotator Cuff Repair Involving Three Tendon Tears
Brief Title: Reverse Shoulder Arthroplasty vs Rotator Cuff Repair for 60+
Acronym: RTSA-RCR
Status: Enrolling by invitation | Type: Observational
Sponsor: Campbell Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-010480-XP
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Injuries; Shoulder Pain
MeSH Terms: conditions — Shoulder Injuries; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reverse Total Shoulder Arthroplasty: Retrospective record review and data abstraction of standard of care data preoperative and at least one year postoperative to include patient reported outcomes and range of motion measurements.
  Interventions: Procedure: Reverse Total Shoulder Arthroplasty
- Rotator Cuff Repair: Retrospective record review and data abstraction of standard of care data preoperative to include patient reported outcomes and range of motion measurements. Study invitation will be extended to subjects for completion of a single study visit to collect three patient reported outcomes, range of motion and a ten minute magnetic resonance imaging exam.
  Interventions: Procedure: Rotator Cuff Repair

INTERVENTIONS:
Procedure: Reverse Total Shoulder Arthroplasty — standard of care treatment reverse total shoulder arthroplasty delivered
  Groups: Reverse Total Shoulder Arthroplasty
Procedure: Rotator Cuff Repair — standard of care treatment rotator cuff repair delivered
  Groups: Rotator Cuff Repair

SUMMARY:
To compare the one year outcomes between 60 year old patients with a three tendon tear treated as part of their standard of care with either a reverse total shoulder arthroplasty or rotator cuff repair surgery.

DETAILED DESCRIPTION:
A retrospective record review will be completed to identify eligible subjects who had either a reverse total shoulder arthroplasty or rotator cuff repair to treat their three tendon tear. Medical record abstraction of standard of care will be completed among the reverse total shoulder arthroplasty cohort. Rotator cuff repair subjects will be contacted with a study invitation and scheduled for a single study visit to collect three patient reported outcomes, assess range of motion and complete a ten-minute magnetic resonance imaging exam following signed consent.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or more at time of surgery
* One year post-reverse total shoulder arthroplasty or one year post-rotator cuff repair involving all three tendons (infraspinatus, supraspinatus, subscapularis)
* Surgery completed by Dr. Tyler Brolin or Dr. Thomas Throckmorton

Exclusion Criteria:

* Less than 60 years of age at time of surgery
* Less than one year post-reverse total shoulder arthroplasty or post-rotator cuff repair
* Procedure completed by another provider than Dr. Brolin or Dr. Throckmorton
* Worker's compensation
* Fewer than three tendon tear

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be patients of either Dr. Brolin or Dr. Throckmorton who had either a reverse total shoulder arthroplasty or rotator cuff repair for treatment of a three tendon tear and are 60 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
American Shoulder Elbow Surgeons | 90 days before surgery to day of surgery
  numeric scale to quantify shoulder function from zero (worst) to one hundred (best)
American Shoulder Elbow Surgeons | one year after surgery
  numeric scale to quantify shoulder function from zero (worst) to one hundred (best)
Visual Analog Scale | 90 days before surgery to day of surgery
  numeric scale to quantify shoulder pain from zero (no pain) to ten (worst pain)
Visual Analog Scale | one year after surgery
  numeric scale to quantify shoulder pain from zero (no pain) to ten (worst pain)
Single Assessment Numeric Evaluation | 90 days before surgery to day of surgery
  Satisfaction with Shoulder
Single Assessment Numeric Evaluation | one year after surgery
  Satisfaction with Shoulder

SECONDARY OUTCOMES:
Revision rate | one year after surgery
  occurrence of repeat surgery
Sugaya | one year after surgery
  Measure of tendon quality from one (intact) to five (completely torn)
Range of motion | 90 day to surgery
  shoulder movement measurement
Range of motion | one year after surgery
  shoulder movement measurement

CONTACTS AND LOCATIONS:
Overall Officials: Tyler J Brolin, MD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared.

REFERENCES:
- [Result] Allert JW, Sellers TR, Simon P, Christmas KN, Patel S, Frankle MA. Massive Rotator Cuff Tears in Patients Older Than Sixty-five: Indications for Cuff Repair versus Reverse Total Shoulder Arthroplasty. Am J Orthop (Belle Mead NJ). 2018 Dec;47(12). doi: 10.12788/ajo.2018.0109. PMID 30650169
- [Result] Jacquot A, Dezaly C, Goetzmann T, Roche O, Sirveaux F, Mole D; French Society for Shoulder, Elbow (SOFEC). Is rotator cuff repair appropriate in patients older than 60 years of age? prospective, randomised trial in 103 patients with a mean four-year follow-up. Orthop Traumatol Surg Res. 2014 Oct;100(6 Suppl):S333-8. doi: 10.1016/j.otsr.2014.04.004. Epub 2014 Aug 23. PMID 25155203
- [Result] Robinson PM, Wilson J, Dalal S, Parker RA, Norburn P, Roy BR. Rotator cuff repair in patients over 70 years of age: early outcomes and risk factors associated with re-tear. Bone Joint J. 2013 Feb;95-B(2):199-205. doi: 10.1302/0301-620X.95B2.30246. PMID 23365029
- [Result] Gowda CS, Mirza K, Galagali DA. Rotator Cuff Tears: Correlation Between Clinical Examination, Magnetic Resonance Imaging and Arthroscopy. Cureus. 2024 Mar 12;16(3):e56065. doi: 10.7759/cureus.56065. eCollection 2024 Mar. PMID 38618461
- [Result] Adam MF, Ladermann A, Denard PJ, Lacerda F, Collin P. Preoperative diagnosis and rotator cuff status impact functional internal rotation following reverse shoulder arthroplasty. J Shoulder Elbow Surg. 2024 Jul;33(7):1570-1576. doi: 10.1016/j.jse.2023.11.020. Epub 2024 Jan 11. PMID 38218405